CLINICAL TRIAL: NCT05638542
Title: Comparison of Expression of Carcinogenesis-related Molecular Markers in the Patients With Colon Cancer and Polyp
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Seoul National University Bundang Hospital (Other)
Responsible Party: Principal Investigator, Nayoung Kim, Professor, Seoul National University Bundang Hospital
Other Study IDs: B-1305-203-009
Record Dates: First submitted 2022-10-26; First posted 2022-12-06 (Actual); Last update posted 2023-04-13 (Actual); Status verified 2023-04

CONDITIONS: Colorectal Cancer; Colorectal Adenoma
Keywords: Carcinogenesis; Sex difference; Tumor location
MeSH Terms: conditions — Colorectal Neoplasms; Carcinogenesis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Endoscopically biopsied samples, blood samples, fecal samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Control group: Patients who are not diagnosed with colorectal adenoma or colorectal cancer
- Colorectal adenoma group: Patients who are diagnosed with colorectal adenoma
- Colorectal cancer group: Patients who are diagnosed with colorectal cancer

SUMMARY:
A study of carcinogenesis-related molecular markers in the patients with colorectal cancer and colorectal adenoma.

DETAILED DESCRIPTION:
The chromosomal instability (CIN) pathway, the CpG island methylator phenotype (CIMP) pathway and the microsatellite instability (MSI) pathway are three major carcinogenesis pathways to colorectal cancer (CRC). In this study, the investigators aimed to investigate distinctive molecular features of carcinogenesis pathways among healthy control, colorectal adenoma, and CRC and compare their molecular progression according to patients' sex and tumor location as well as disease stage.

ELIGIBILITY:
Inclusion Criteria:

* Control group: subjects with no evidence of colorectal adenoma or colorectal cancer
* Colorectal adenoma group: Patients with colorectal adenomas greater than or equal to 10 mm in diameter according to the endoscopic presentation as well as histological validation of colorectal adenoma.
* Colorectal cancer group: Patients whose biopsy specimen is histologically confirmed as colorectal adenocarcinoma

Exclusion Criteria:

* Subjects age under 18 years
* Previous history of colorectal neoplasms
* Patients with high bleeding risk or patients who must maintain anti-coagulant or anti-platelet agents
* Denial to participate in this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients who visited Seoul National University Bundang Hospital for gastrointestinal symptomes or regular check-ups, and agreed to participate.
Sampling Method: Non-Probability Sample
Enrollment: 582 (Actual)
Dates: Start 2015-03-01 (Actual); Primary Completion 2021-01-30 (Actual); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
The characteristics of carcinogenesis-related molecular markers in colorectal adenoma and CRC | through study completion, an average of 1 year
  Using endoscopically biopsied specimens, multiple carcinogenic markers were investigated including KRAS and BRAF mutation, PD-L1, EGFR, IL-1b, NLRP3, Caspase-1, p53 expression, Microinstability (MSS, MSI-L, MSI-H), PD-L1, DNA mismatch repair proteins (MLH1, MSH2, MSH6, PMS2), CIMP markers (p16, MINT1, MINT2, MINT31, hMLH1), promoter methylation of p16, RUNX3, NEUROG1.
  CIMP was assessed by methylation-specific PCR for five methylation panel markers (p16, MINT1, MINT2, MINT31, hMLH1), and MSI status was validated by PCR using five NCI markers (BAT-26, BAT-25, D5S346, D17S250, and S2S123). KRAS and BRAF mutation was analyzed by direct sequencing using sequence-specific primers from the acquired biopsy specimens. PD-L1, EGFR, MMR expression was examined using immunohistochemistry.
Fecal microbiota analysis in patients with colorectal adenoma and CRC | through study completion, an average of 1 year
  Using next-generation sequencing technique, fecal microbiota of patients with colorectal adenoma and CRC as well as healthy control was evaluated to verify carcinogenesis-related microbiota.

CONTACTS AND LOCATIONS:
Overall Officials: Nayoung Kim, M.D., Ph.D, Study Chair — Seoul National University Bundang Hospital
Locations (1):
- Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Choi J, Kim N, Nam RH, Kim JW, Song CH, Na HY, Kang GH. Influence of location-dependent sex difference on PD-L1, MMR/MSI, and EGFR in colorectal carcinogenesis. PLoS One. 2023 Feb 21;18(2):e0282017. doi: 10.1371/journal.pone.0282017. eCollection 2023. PMID 36802389